CLINICAL TRIAL: NCT06144281
Title: Study of Home-Embedded Palliative Care for Hemodialysis- (and Peritoneal-) Dependent End-Stage Renal Disease (SHEPHERD 2.0)
Brief Title: Study of Home-Embedded Palliative Care for Hemodialysis- (and Peritoneal-) Dependent End-Stage Renal Disease
Acronym: SHEPHERD 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Effectiveness of home palliative care services could not be determined due to lower-than-expected referrals and consults in the intervention arm
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 851328 (2)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: End-Stage Renal Disease
Keywords: palliative; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The inpatient care team, including the attending/ordering and covering providers, for participants in this group will receive a message from the research team identifying their patient as appropriate for home palliative care and will be asked to refer their patient for these services.
  Interventions: Behavioral: Nudge for PHPC NP Referral
- Usual Care (No Intervention): Participants in this group will receive usual care upon discharge from the hospital. Their clinical team will not be notified that they are appropriate for home palliative care services, but they may still be referred for those services if their clinicians feel their patient will benefit.

INTERVENTIONS:
Behavioral: Nudge for PHPC NP Referral — The attending and covering providers for inpatients who have been identified according to the study's inclusion criteria as appropriate for home palliative care services upon hospital discharge will be asked to refer their patient for these services.
  Arms: Intervention

SUMMARY:
Home palliative care needs are often under-recognized in patients with End-Stage Renal Disease (ESRD). This pilot study is designed to evaluate the effectiveness of referrals to home palliative care services in improving patient outcomes compared with usual care among patients with ESRD admitted to a Penn hospital. Evaluating the effectiveness of home palliative care services is critical to determine whether increasing access to these services would improve patient-centered outcomes for these high-need patients

ELIGIBILITY:
Inclusion Criteria:

* Be an adult (18 years of age or older) hospitalized at a Penn study hospital
* AND digital signature of ESRD (N18.6) within the last 12 months
* AND resides in the five-county area surrounding Philadelphia which is served by Penn Palliative Care Nurse Practitioner program
* AND have one or more of the following markers of potentially unmet needs: (i) existing home care eligibility or referral for home care (but not already receiving PC); (ii) non-ambulatory status determined via nursing assessment; (iii) severe protein-calorie malnutrition; (iv) 2 or more hospitalizations within the prior year

Exclusion Criteria:

* Patients with functional kidney transplants
* Patients discharged to skilled nursing facilities and LTC facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Acute Encounters | Baseline - 180 days
  A combined count of hospitalizations, Emergency Department, and Observation visits during the 180-day follow-up period that will be assessed using the electronic health record and administrative data for the tri-state area

SECONDARY OUTCOMES:
Hospital-Free Days | Baseline - 180 days
  The number of hospital-free days during the 180-day follow-up period will be assessed using the electronic health record and administrative data for the tri-state area.
Home Palliative Care Visits | Baseline - 180 days
  The total number of home palliative care visits during the 180-day follow-up period after hospital discharge will be assessed using the electronic health record.
Time to Home Palliative Care Visit | Baseline - 180 days
  Days from hospital discharge to the first home palliative care visit.
Mortality | Baseline - 180 days
  Mortality rates will be assessed using the electronic health record after the 180-day follow-up period.
Hospice Enrollment | Baseline - 180 days
  New hospice enrollment will be assessed using the electronic health record and administrative data for the tristate area.
Health-Related Quality of Life | 1- and 3-months
  Health-related quality of life will be assessed by the EQ-5D survey of patients at 1- and 3-months post-hospital discharge time-points.
Symptom Burden | 1- and 3-months
  Symptom burden will be assessed by the Edmonton Symptom Assessment System survey of patients at 1- and 3-months post-hospital discharge time-points.
Quality of Care | 1- and 3-months
  Quality of care will be assessed by the CMS-MACRA PC Quality Measures (Received Help for Pain; Felt Heard & Understood) for patients at 1- and 3-months post-hospital discharge time-points.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States